CLINICAL TRIAL: NCT05575895
Title: Evaluation of Systemic Microvascular Reactivity After Ingestion of an Energy Drink in Young Male Volunteers
Status: Completed | Type: Observational
Sponsor: National Institute of Cardiology, Laranjeiras, Brazil (Other Government)
Responsible Party: Principal Investigator, Eduardo Tibirica, MD, PhD, Senior researcher, National Institute of Cardiology, Laranjeiras, Brazil
Other Study IDs: CAAE 13135219.0.0000.5272
Record Dates: First submitted 2022-10-05; First posted 2022-10-12 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Endothelial Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Energy Drink: Ingestion of 250 ml of the energy drink (Red Bull®)
  - Evaluation of systemic skin microvascular endothelial function Laser-based method for evaluating non-invasive, operator-independent systemic microvascular function that detects microvascular flow in the skin for the evaluation of systemic vascular endothelial function.
  Interventions: Dietary Supplement: Ingestion of the energy drink (Red Bull®)
- Control: Ingestion of 250 ml of mineral water (Minalba®)
  - Evaluation of systemic skin microvascular endothelial function Laser-based method for evaluating non-invasive, operator-independent systemic microvascular function that detects microvascular flow in the skin for the evaluation of systemic vascular endothelial function.
  Interventions: Dietary Supplement: Ingestion of mineral water

INTERVENTIONS:
Dietary Supplement: Ingestion of the energy drink (Red Bull®) — Ingestion of 250 ml of the energy drink (Red Bull®)
  Groups: Energy Drink
Dietary Supplement: Ingestion of mineral water — Ingestion of 250 ml of mineral water (Minalba®)
  Groups: Control

SUMMARY:
Purpose: Energy drinks (EDs) are nonalcoholic beverages whose main ingredients are sugar, taurine, and caffeine. Their consumption is rising worldwide, with only few conflicting studies examining their vascular effects in young adults. We evaluated microvascular reactivity (MR) before and after ED in young healthy male volunteers.

Methods: Systemic MR was evaluated in the skin of the forearm using laser speckle contrast imaging with acetylcholine (ACh) iontophoresis before, 90 and 180 minutes after the consumption of one can of ED or the same volume of water (control), followed by postocclusive reactive hyperemia (PORH).

DETAILED DESCRIPTION:
Energy drinks (EDs) are nonalcoholic beverages whose main ingredients are sugar, taurine, and caffeine. These products are marketed as boosters of mental and physical performance and are increasingly used in Western societies. Case reports of adverse effects related to ED consumption have been described in healthy young individuals, including coronary artery vasospasm, and myocardial infarction. These data suggest that endothelial dysfunction (EDysf) plays a role in ED cardiovascular effects and have prompted studies with conflicting results. The present study evaluated the microvascular reactivity (MR) after ingestion of one can of ED compared to a control, in young healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* healthy male volunteers with no relevant findings in the medical history

Exclusion Criteria:

* being a competitive athlete;
* being on regular medication;
* using illicit drugs;
* being allergic to coffee, taurine or any of the components of the selected energy drink; - -
* having a body mass index ≥ 30 kg/m2.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy male volunteers with no relevant findings in the medical history
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Endothelium-dependent skin microvascular reactivity | Microvascular reactivity will be evaluated after a 20-minute rest in the supine position in a temperature-controlled room.
  Cutaneous microvascular flow measured with laser speckle contrast imaging

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - National Institute of Cardiology, Ministry of Health, Brazil, Rio de Janeiro
  - Eduardo Tibiriçá, Rio de Janeiro